CLINICAL TRIAL: NCT01962584
Title: Value of CMR Including T1 Mapping in Patients With Acute Myocarditis
Brief Title: CMR in Patients With Myocarditis
Status: Completed | Type: Observational
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Claas P. Naehle, section chief cardicvascular imaging, University Hospital, Bonn
Other Study IDs: 150/13
Record Dates: First submitted 2013-10-04; First posted 2013-10-14 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Suspected Acute Myocarditis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- SAM: patients with suspected acute myocarditis
- HC: Healthy controls

SUMMARY:
To evaluate the additive values of T1 mapping in patients with acute myocarditis.

DETAILED DESCRIPTION:
Cardiac magnetic resonance (CMR) is an established non-invasive diagnostic tool for acute and chronic myocarditis. Established CMR criteria for diagnosing myocarditis are edema on black-blood T2-weighted imaging, relative contrast enhancement seen on T1-weighted imaging for assessment of hyperemia, and late contrast-agent enhancement seen with inversion recovery late enhancement technique for visualization of myocardial fibrosis.

Recently, tissue characterization based on calculation of myocardial T1 relaxation time (T1 mapping) as well as T1-derived extracellular volume fraction has become available. Recently, reference values for myocardial T1 relaxation times at 3T for healthy volunteers were published for CMR. However, to date no comprehensive data for multiparametric CMR in patients with suspected myocarditis at 3 Tesla is available. Therefore, the purpose of this prospective study was to evaluate the diagnostic value of CMR at 3T in patients with suspected acute myocarditis using a multiparametric CMR approach including T1 mapping as novel tool for tissue characterization.

CMR will be performed within 7 days after hospital admission for "suspected acute myocarditis".

ELIGIBILITY:
Inclusion Criteria:

* patients with suspected acute myocarditis and otherwise unremarkable cardiac history

Exclusion Criteria:

* exclusion of CAD in invasive coronary angiography
* pregnancy
* contraindications for MR imaging

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: patients with suspected acute myocarditis and otherwise unremarkable cardiac history exclusion of CAD in invasive coronary angiography
Sampling Method: Non-Probability Sample
Enrollment: 66 (Actual)
Dates: Start 2013-09; Primary Completion 2014-10 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
T1 relaxation times | time of CMR, CMR will be performed within 7 days after hospital admission for "suspected acute myocardtitis".
  quantification of T1 relaxation times

SECONDARY OUTCOMES:
Extracellular volume (ECV) | time of CMR, CMR will be performed within 7 days after hospital admission for "suspected acute myocardtitis".
  calculation of extracellular volume based on T1 relaxation time

CONTACTS AND LOCATIONS:
Locations (1):
- University of Bonn, Bonn, North Rhine-Westphalia, Germany